CLINICAL TRIAL: NCT04965584
Title: A Study Focused on the Microflora and Metabolomics of Crohn's Disease Patients
Brief Title: Microflora and Metabolomics of Crohn's Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Professor, Shanghai 10th People's Hospital
Other Study IDs: SHSYXK
Record Dates: First submitted 2021-07-12; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; microbiota; metabonomics
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active Crohn's disease group: Patients diagnosed with Crohn's disease after comprehensive evaluation of clinical symptoms, endoscopic features, radiological manifestations and histological features were recruited, and patients with CDAI score ≥ 150 were included in this group.
- Crohn's disease remission group: Patients diagnosed with Crohn's disease after comprehensive evaluation of clinical symptoms, endoscopic features, radiological features and histological features were recruited, and patients with CDAI score < 150 were included in this group.
- Healthy control group: Normal healthy people were randomly recruited as the control group

SUMMARY:
The purpose of this study is to explore the microflora characteristics of different ecological loci and multiple metabolic pathways in Crohn's disease patients with different disease course states.

DETAILED DESCRIPTION:
This study aims to investigate the characteristics of microflora in the oral and tongue base, small intestinal stomy and lower respiratory tract, as well as the characteristics of multiple metabolic pathways such as bile acid metabolism and amino acid metabolism in Crohn's disease patients with different course states.

ELIGIBILITY:
Inclusion Criteria:

1. individuals who were clear and signed the informed consent.
2. Male and female.

Exclusion Criteria:

1. Any one who can not provide accurate information.
2. Any one who denies the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three different groups were created by healthy volunteers, patients with active Crohn's disease and patients with remission of Crohn's disease. The information of these individuals will be analyzed and some conclusions will be drawn.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Oral microbiota structure and function difference between active stage of Crohn's disease, remission of Crohn's disease and healthy controls | 3 months
  The results were based on the 16S rRNA sequencing
Small intestinal microbiota structure and function difference between active stage of Crohn's disease, remission of Crohn's disease and healthy controls | 3 months
  The results were based on the 16S rRNA sequencing
Sputum microbiota structure and function difference between active stage of Crohn's disease, remission of Crohn's disease and healthy controls | 3 months
  The results were based on the 16S rRNA sequencing

SECONDARY OUTCOMES:
Metabolic difference of blood samples between active stage of Crohn's disease, remission of Crohn's disease and healthy controls | 3 months
  The metabolites of the blood samples by LC-MS will be detected

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xia K, Gao R, Wu X, Sun J, Wan J, Wu T, Fichna J, Yin L, Chen C. Characterization of Specific Signatures of the Oral Cavity, Sputum, and Ileum Microbiota in Patients With Crohn's Disease. Front Cell Infect Microbiol. 2022 Apr 13;12:864944. doi: 10.3389/fcimb.2022.864944. eCollection 2022. PMID 35493739